CLINICAL TRIAL: NCT04104399
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Single Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of XC101-D13H in Healthy Adult Subjects
Brief Title: Single Ascending Dose Study to Investigate the Safety and Pharmacokinetics of XC101-D13H in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xoc Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XC101-D13H-CL-1
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XC101-D13H (Experimental): single dose
  Interventions: Drug: XC101-D13H
- Placebo (Placebo Comparator): single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC101-D13H — XC101-D13H supplied as 0.4, 0.8, 1.6 or 3.2 mg dose, administered in capsules
  Arms: XC101-D13H
Drug: Placebo — Placebo supplied as matching capsules
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group single ascending dose (SAD) study. There are 4 cohorts of 8 subjects (8 active and 2 placebo) planned for evaluation under fasting conditions. One of the planned dose levels will cross over after a washout period to receive the same single dose of XC101-D13H or placebo under fed conditions.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group single ascending dose (SAD) study. There are 4 cohorts of 8 subjects (8 active and 2 placebo) planned for evaluation under fasting conditions. One of the planned dose levels will cross over after a washout period to receive the same single dose of XC101-D13H or placebo under fed conditions. Dose escalation will be supervised by a Safety Monitoring Board (SMB). Dose escalation to the next dose level will not take place until the SMB has determined that adequate safety, tolerability, PK, and core-lab analyzed ECGs from the previous cohort and all previous cohorts have been demonstrated to permit proceeding to the next cohort. PK data from all available cohorts will be used to guide the dose-escalation decisions.

ELIGIBILITY:
Major Inclusion Criteria:

* Healthy, adult, male or female of non childbearing potential only, 18-55 years of age, inclusive, at screening.
* Body mass index (BMI) ≥ 18 and ≤ 30.0 kg/m2 at screening.
* Medically healthy with no clinically significant finding in medical history, physical examination, laboratory profiles, vital signs, or ECGs, as judged by the PI or designee. Creatinine must be within the upper limit of normal at screening.
* Understands the study procedures in the informed consent form (ICF), and is willing and able to comply with the protocol.

Major Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical, surgical, clinical laboratory, or psychiatric condition or disease.
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* History of clinically significant hypotension.
* History of lightheadedness, dizziness or syncope in the 12 months prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2022-01-28 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | pre-dose through 14 days post-dose
  Adverse Events will be monitored throughout confinement in the clinic and through the 14-day follow-up visit.

SECONDARY OUTCOMES:
Maximum plasma concentration [Cmax] of XC101-D13H | 48 hours
  Blood samples will be collected pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose and the maximum observed concentration for XC101-D13H will be calculated.
Area under the curve [AUC] of XC101-D13H | 48 hours
  Blood samples will be collected pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose and the area under the concentration-time curve, from time 0 to the last observed non-zero concentration will be calculated for XC101-D13H.
Time to reach maximum plasma concentration [Tmax] of XC101-D13H | 48 hours
  Blood samples will be collected pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose and the time to reach the maximum plasma concentration of XC101-D13H will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fishman, MD, Study Director — Xoc Consulting Chief Medical Officer
Locations (1):
- Celerion, Tempe, Arizona, United States